CLINICAL TRIAL: NCT02864225
Title: A Prospective, Blinded Clinical Study to Compare the Efficacy Between Three Fetal Monitoring Methods: Electro Uterine Monitor (EUM), Fetal Doppler and Scalp Electrode
Brief Title: To Compare the Efficacy Between 3 Fetal Monitoring Methods (EUM)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: 573-15-TLV
Record Dates: First submitted 2016-08-08; First posted 2016-08-11 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-08

CONDITIONS: Fetal Heartbeat Tracings

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Scalp electrode, fetal doppler and EUM (Experimental): Once in labor, the parturient will be connected to the routine fetal doppler and EUM. When necessary according to clinical indications, the scalp electrode will be connected. Tracing will be recorded simultaneously from all three devices until delivery.
  Interventions: Device: Scalp electrode,; Device: Fetal doppler; Device: EUM

INTERVENTIONS:
Device: Scalp electrode, — the parturient will be connected to the routine fetal Doppler and to the EUM. and When necessary to the scalp electrode will be connected. Tracings will be recorded simultaneously from all three devices until delivery. three separate outputs will be processed Output of the scalp electrode recording. Output of the fetal doppler. Output of the EUM. Three noncontinuous segments of 30 minutes each with two segments occurring during the first stage of labor and the third occurring during the second stage of labor, will be randomly picked from the scalp electrode recording with 3 matching segments in time from the EUM100pro and the fetal doppler
Device: Fetal doppler — the parturient will be connected to the routine fetal Doppler and to the EUM. and When necessary to the scalp electrode will be connected. Tracings will be recorded simultaneously from all three devices until delivery. three separate outputs will be processed Output of the scalp electrode recording. Output of the fetal doppler. Output of the EUM. Three noncontinuous segments of 30 minutes each with two segments occurring during the first stage of labor and the third occurring during the second stage of labor, will be randomly picked from the scalp electrode recording with 3 matching segments in time from the EUM100pro and the fetal doppler
Device: EUM — the parturient will be connected to the routine fetal Doppler and to the EUM. and When necessary to the scalp electrode will be connected. Tracings will be recorded simultaneously from all three devices until delivery. three separate outputs will be processed Output of the scalp electrode recording. Output of the fetal doppler. Output of the EUM. Three noncontinuous segments of 30 minutes each with two segments occurring during the first stage of labor and the third occurring during the second stage of labor, will be randomly picked from the scalp electrode recording with 3 matching segments in time from the EUM100pro and the fetal doppler

SUMMARY:
Background:

Identification and measurement of fetal heart tracings throughout pregnancy and labor is crucial to the well-being of the fetus. Non reassuring fetal heart rate is one of the most common indications for operative vaginal delivery or cesarean section. Therefore, management of labor requires reliable and accurate information about fetal heart rate.

In most normal spontaneous labors, fetal heart rate is characterized by the baseline heart rate (from 110 to 160 beats per minute), variability (beat to beat changes) and periodic changes (accelerations or decelerations). In each stage of labor the tracing may have different characteristics, with variable decelerations much more common at the end of the second stage of labor.

Objective:

To Show non inferiority of the EUM to the fetal doppler and scalp electrode by comparing the reliability and accuracy of the EUM versus fetal doppler compared to scalp electrode in the same patients.

DETAILED DESCRIPTION:
Background:

Identification and measurement of fetal heart tracings throughout pregnancy and labor is crucial to the well-being of the fetus. Non reassuring fetal heart rate is one of the most common indications for operative vaginal delivery or cesarean section. Therefore, management of labor requires reliable and accurate information about fetal heart rate.

In most normal spontaneous labors, fetal heart rate is characterized by the baseline heart rate (from 110 to 160 beats per minute), variability (beat to beat changes) and periodic changes (accelerations or decelerations). In each stage of labor the tracing may have different characteristics, with variable decelerations much more common at the end of the second stage of labor.

Objective:

To Show non inferiority of the EUM to the fetal doppler and scalp electrode by comparing the reliability and accuracy of the EUM versus fetal doppler compared to scalp electrode in the same patients.

METHODS The current method for detecting fetal heart rate is fetal Doppler, which is routinely used in practically all labors, is based on the Doppler technology of detecting heart valves motion and blood velocity. The fetal Doppler transducer is placed on the abdomen of the parturient and is susceptible to positional changes of the parturient. Moreover, among obese gravidas, fetal heart rate tracings via external fetal Doppler may be difficult to achieve.

Another method for monitoring fetal heart rate is the scalp electrode which is attached to the fetal scalp and records the heart rate patterns. This method is invasive and can be used only after the amniotic membranes are ruptured.

Monitoring with scalp electrode is superior to the fetal Doppler as it is direct and non-affected by maternal position. However, it is an invasive method and may contribute to the development fever during or after labor.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical indication to insert a scalp electrode for fetal heart rate tracing.
2. Maternal age >18 years
3. Reactive fetal heart rate monitoring and BPP 8/8 at enrollment
4. Singleton pregnancy
5. No fetal abnormality or chromosomal defect
6. Subjects are willing and able to comply with the requirements of the protocol.
7. Fully understand all elements of, and have signed and dated, the written informed consent form before initiation of protocol-specified procedures, when VAS <3.

Exclusion Criteria:

1. Women who refused to sign the informed consent form.
2. Maternal age < 18 years.
3. Multiple pregnancy
4. Woman with implanted electronic device of any kind
5. Woman with allergic to silver.
6. Irritated skin or open wound

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2016-09; Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
The difference between the fetal scalp electrode tracings and the EUM tracings of the fetal heart activity. | Up to 72 hours
  Mean Positive Percent Agreement (PPA) for interpretable/un interpretable traces (between EUM, scalp electrode and fetal doppler).
Reliability | Up to 72 hours
  Mean sensitivity for individual tracing identification (between EUM, scalp electrode and fetal doppler)
Reliability | Up to 72 hours
  Mean Positive Predictive Value (PPV) for individual tracing identification (between EUM, scalp electrode and fetal doppler)
Reliability | Up to 72 hours
  The mean False Positive Rate (FPR) for individual tracing identification (between EUM, scalp electrode and fetal Doppler)

CONTACTS AND LOCATIONS:
Overall Officials: Yariv Yogev, professor, Study Chair — Tel Aviv Medical Center

IPD SHARING:
Plan to Share IPD: No